CLINICAL TRIAL: NCT06498791
Title: Functional Mitochondrial Analysis of Peripheral Blood Mononuclear Cells (PBMCs) - a Pilot Study
Brief Title: Functional Mitochondrial Analysis PBMCs
Acronym: FMAP
Status: Active, not recruiting | Type: Observational
Sponsor: VASCage GmbH (Other)
Collaborators: Oroboros Instruments (Unknown)
Responsible Party: Sponsor
Other Study IDs: C_2_A.7-0039_009
Record Dates: First submitted 2024-06-18; First posted 2024-07-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mitochondrial Function
Keywords: Mitochondrial respiration; PBMC
MeSH Terms: interventions — Phlebotomy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Venipuncture — Blood drawing
Other: Questionnaire — Completion of the questionnaire

SUMMARY:
The primary goal of this prospective, exploratory, longitudinal, single-centre, cohort study is to assess the stability of the mitochondrial flux in PBMCs over long-term cryopreservation.

Secondary goals of this study are:

* to identify changes in the mitochondrial respiratory flux in different metabolic states of cryopreserved PBMCs during long-term cryopreservation.
* to assess variability between mitochondrial respiration from PBMCs isolated from same volunteers at different times, seasons or from different arms.

DETAILED DESCRIPTION:
The analysis of mitochondrial function can also be referred to as a bioenergetic snapshot. Mitochondria are dynamic metabolic organelles that adapt to various physiological demands, reflecting an individual's lifestyle and exposure to environmental factors, medications, and toxins. Numerous studies have shown that mitochondrial respiration declines with age and correlates with many age-related diseases. This raises the question of how mitochondria influence cells in a clinical context.

For this purpose, 20 participants are recruited and comprehensively characterized in terms of their demographic information and clinical profiles. Additionally, physical examinations are conducted, and participants are surveyed about their lifestyles through questionnaires. Over a 12-month period, blood samples are collected at intervals of three months, resulting in a total of five study visits. For the analysis of mitochondrial oxygen consumption, peripheral blood mononuclear cells (PBMCs) are preferably used, as they provide a minimally invasive and easily accessible insight into mitochondrial function and overall metabolic status and are isolated from the collected blood samples.

To enable the application of mitochondrial diagnostics in research for early disease detection and therapeutic development, additional information is needed regarding the stability of mitochondrial respiration in cryopreserved PBMCs using high-resolution respirometry (HRR) with O2k technology. The goal of this study is to assess how the duration of cryopreservation affects mitochondrial bioenergetics compared to freshly isolated PBMCs.

The study also considers a variety of parameters that could potentially influence the stability of mitochondrial respiration. These factors include non-fasting blood collection, discrepancies between the right and left arm, and seasonal effects. To what extent the intraindividual variability in these parameters affects the mitochondrial respiration is yet to be fully understood.

Furthermore, the longitudinal study design allows the tracking of mitochondrial activity and stability over time, providing a better understanding of the central processes of cellular respiration.

Thus, the planned study promises to yield significant insights into mitochondrial respiration and cellular bioenergetics in a clinical context.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-85
* Willingness and ability to consent

Exclusion Criteria:

* Regular (e.g. daily, weekly or similar) intake of medication or nutritional supplements except oral and spiral contraceptives
* Autoimmune diseases or immune alterations
* Diseases in the context of haematopoiesis, haemophilia, hematophobia
* Diagnosed mild or major neurocognitive disorder
* Depressive episodes in the last two years
* Chronic infectious diseases
* Neurostimulators or drug pump
* Involved in competitive sports (over the past two years)
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The source population for this study comprises adults (older than 18 years of age) with an equal distribution of male and female.
  Overall, 20 individuals will be included in the study (10 male, 10 female).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Stability of mitochondrial respiratory flux (O2 flux) in cryopreserved PBMCs | 1 week and every 8 weeks after cryopreservation
  Mitochondrial respiratory flux is assessed by High Resolution Respirometry analysis
Stability of O2 concentration in cryopreserved PBMCs | 1 week and every 8 weeks after cryopreservation
  Mitochondrial respiratory flux is assessed by High Resolution Respirometry analysis
Assessment of mitochondrial respiratory flux (O2 flux) in fresh PBMCs compared to cryopreserved PBMCs | Baseline visit, 3, 6, 9, 12 months visit
  Mitochondrial respiratory flux is assessed by High Resolution Respirometry analysis
Assessment of O2 concentration in fresh PBMCs compared to cryopreserved PBMCs | Baseline visit, 3, 6, 9, 12 months visit
  Mitochondrial respiratory flux is assessed by High Resolution Respirometry analysis

SECONDARY OUTCOMES:
Assessment of O2 flux in fresh and cryopreserved PBMCs in fasted vs non-fasted sampling conditions | 6 months visit
  Assessement of mitochondrial bioenergetic snapshot in fresh and cryopreserved PBMCs at two different collection time points (fasted and non-fasted)
Assessment of O2 flux in fresh and cryopreserved PBMCs at different seasonal collection time points | Baseline visit, 3, 6, 9, 12 months visit
  Assessement of mitochondrial bioenergetic snapshot in fresh and cryopreserved PBMCs in different seasons
Assessment of O2 flux in fresh and cryopreserved PBMCs at different venipuncture sites | 3 months visit
  Assessement of mitochondrial bioenergetic snapshot in fresh and cryopreserved PBMCs collected from left and right arm
Assessment of blood count and differential blood count I | Baseline visit, 3, 6, 9, 12 months visit
  Analysis of complete blood count (e.g. erythrocyte concentration (mg/dL))
Assessment of blood count and differential blood count II | Baseline visit, 3, 6, 9, 12 months visit
  Analysis of complete blood count (e.g. haemoglobin concentration (g/dL))
Concentration of Creatinine and Urea | Baseline visit, 3, 6, 9, 12 months visit
  Creatinine (mg/dL), Urea (mg/dL)
Concentration of Creatine Kinase | Baseline, 6, 12 months visit
  Creatine Kinase (U/L)
Concentration of Glucose | Baseline visit, 3, 6, 9, 12 months visit
  Glucose (mg/dL, mmol/L)
Concentration of HbA1c | Baseline, 6, 12 months visit
  HbA1c (%)
Concentration of Sodium, Potassium, Chloride and Calcium | Baseline, 6, 12 months visit
  Sodium (mmol/L), potassium (mmol/L), chloride (mmol/L), calcium (mmol/L)
Concentration of GOT and GPT | Baseline, 6, 12 months visit
  Glutamic-oxaloacetic transaminase (GOT, U/L), glutamic-pyruvic transaminase (GPT, U/L), gamma-glutamyl-transpeptidase (gamma-GT, U/L), lactate dehydrogenase (LDH, U/L)
Concentration of triglyceride and cholesterol | Baseline, 6, 12 months visit
  Triglyceride (mmol/L), cholesterol (all, mmol/L )
Concentration of LDL-cholesterol and HDL-cholesterol | Baseline, 6, 12 months visit
  LDL-cholesterol (mg/dL), HDL-cholesterol (mg/dL)
Concentration of Lipoprotein a | Baseline visit
  Lipoprotein a (mg/dL)
Assessment of Sedimentation rate | Baseline, 12 months visit
  Sedimentation rate (mm/h)
Concentration of C-reactive protein | Baseline visit, 3, 6, 9, 12 months visit
  CRP sensitive (mg/L)
Concentration of Interleukin-6 | Baseline, 6, 12 months visit
  Interleukin-6 (pg/ml)
Concentration of Thyroid-stimulating hormone | Baseline, 12 months visit
  TSH (mU/mL)
Concentration of Iric acid | Baseline, 12 months visit
  Uric acid (mg/dL)
Concentration of Ferritin | Baseline, 12 months visit
  Ferritin (ng/mL, μg/L)

OTHER OUTCOMES:
Demographic data I | Baseline visit
  Assessment of demographic data such as current age, sex at birth, location of birth
Demographic data II | Baseline visit
  Assessment of demographic data such as: height (cm)
Demographic data III | Baseline visit
  Assessment of demographic data such as: weight (kg)
Demographic data - Personal background and lifestyle I | Baseline visit
  Assessment of demographic data with focus on personal background and lifestyle: e.g.
  * ethnicity (anamnesis)
  * marital/relationship status (anamnesis)
  * number of children (anamnesis)
  * highest level of education (anamnesis)
Menstrual cycle duration (women only) | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of menstrual cycle with focus on cycle duration (in days)
Menstrual cycle length (women only) | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of menstrual cycle with focus on the initiation of the last cycle (day)
Demographic data - Personal background and lifestyle II | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of demographic data with focus on personal background and lifestyle: smoking and smoking history, alcohol consumption and diet
Demographic data - Personal background and lifestyle III | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of demographic data with focus on personal background and lifestyle: amount and intensity of physical activity
Demographic data - Personal background and lifestyle IV | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of personal background and lifestyle: sleep quality
Medical History Assessment | Baseline visit, 3, 6, 9, 12 months visit
  Assessment of medical history:
  * pre-existing illnesses
  * current illnesses or allergies
  * chronic illnesses
  * medication
  * previous surgical procedures within the last 2 years
Assessment of mental well-being using the Hospital Anxiety and Depression Scale - German Version (HADS-D) questionnaire | Baseline visit, 3, 6, 9, 12 months visit
  The questionnaire uses an anxiety scale and a depression scale (0-21, each). The higher the value, the more anxious/depressed the patient. Cut-off for clinical significance: ≥8

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, AssozProf Dr, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University Innsbruck - Department of Neurology, Innsbruck, Tyrol, Austria